CLINICAL TRIAL: NCT06450639
Title: A Phase II Multicenter, Open-label Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Satralizumab in Pediatric Patients With Duchenne Muscular Dystrophy (SHIELD DMD)
Brief Title: A Study to Assess the Efficacy and Safety of Satralizumab in Duchenne Muscular Dystrophy (DMD)
Acronym: SHIELD DMD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN45398; 2024-512383-65-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD, IL6, IL6R, bone, muscle, fractures, BMD, inflammation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Fractures, Bone; Inflammation | interventions — satralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Satralizumab (Experimental): Participants will receive satralizumab SC injection on Day 1, Weeks 2 and 4 (loading doses) and then Q4W from Weeks 8 to 104 (maintenance doses) until the study completion visit.
  Interventions: Drug: Satralizumab

INTERVENTIONS:
Drug: Satralizumab — Satralizumab will be administered SC in the abdominal or femoral region on Day 1, Weeks 2 and 4 (loading doses) and then Q4W from Weeks 8 to 104 (maintenance doses) until the study completion visit.

SUMMARY:
The purpose of this study is to assess the efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of satralizumab, a humanized anti-interleukin-6 receptor (aIL-6R) monoclonal antibody, in ambulatory and non-ambulatory participants with DMD age ≥ 8 to < 18 years old receiving corticosteroid therapy.

DETAILED DESCRIPTION:
Participants will be included in two groups: ambulatory participants with fractures and non-ambulatory participants with or without a history of fractures (Group 1) and ambulatory participants who are fracture naive (Group 2) at baseline. The study will assess the potential of satralizumab to improve bone fragility and to increase muscle function. A weight tier based dose of satralizumab will be given by subcutaneous (SC) injection every 4 weeks (Q4W).

ELIGIBILITY:
Key Inclusion Criteria:

* Signed Informed Consent Form and Signed Assent Form when appropriate
* Male at birth
* A definitive diagnosis of DMD prior to screening based on documentation of clinical findings and prior confirmatory genetic testing using a clinical diagnostic genetic test
* Age ≥ 8 and < 18 years at the time of signing Informed Consent Form
* Group 1 participants are required to meet the following criteria:

  - Ambulatory (defined as able to walk independently without assistive devices) with a prior history of fractures:
  1. Prior history of low-trauma fracture defined as: evidence of at least one prevalent vertebral compression fracture of Genant Grade 1 or 2 (or radiographic signs of VF) or history of at least one low-trauma long-bone fracture (upper or lower extremity) OR
  2. Non-ambulatory, characterized as being non-ambulatory for a minimum of 6 months with onset of non-ambulatory status defined as participant- or caregiver-reported age of continuous wheelchair use approximated to the nearest month, and an North Star Ambulatory Assessment (NSAA) walk score of "0" and inability to perform the 10-Meter Walk/Run (10 MWR) at the baseline visit, with or without fractures
* Group 2 participants are required to meet the following criteria:

  * Be fracture naïve, defined as: no history of prior low-trauma fractures before the baseline visit nor any radiological findings indicative of prevalent VF at the screening visit
  * Be ambulatory defined as able to walk independently without assistive devices
  * Age ≥ 8 to < 12 years old at the time of screening
* Daily oral corticosteroids

Key Exclusion Criteria:

* Major surgery (e.g. spinal surgery) within 3 months prior to Baseline or planned surgery or procedure that would interfere with the conduct of the study for any time during this study
* Presence of any clinically significant illness
* Has serological evidence of current, chronic, or active human immunodeficiency virus (HIV), tuberculosis (TB), hepatitis C, or hepatitis B infection
* Has a symptomatic infection (e.g. upper respiratory tract infection, pneumonia, pyelonephritis, meningitis) within 4 weeks prior to baseline
* Body weight at screening <20 or > 100 kg
* Evidence of a severe vertebral fracture (VF) (defined as Grade 3), assessed by radiographic imaging at screening and quantified using the Genant semiquantitative method
* Treatment with prohibited therapies as defined by the protocol
* Has received a live or live attenuated virus vaccine within 6 weeks of the Baseline visit or expects to receive a vaccination during the first 3 months after Baseline.
* Has abnormal laboratory values considered clinically significant as defined by the protocol
* Any medical condition that might interfere with the evaluation of LS BMD, such as severe scoliosis or spinal fusion.
* Participant has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the investigator
* Participant has an allergy or hypersensitivity to the study medication or to any of its constituents

Other protocol defined inclusion and exclusion criteria may apply

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male participants
Enrollment: 50 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Group 2: Change From Baseline to Week 52 in Lumbar Spine (LS) Bone Mineral Density (BMD) Z-score Measured by Dual-energy X-ray Absorptiometry (DEXA) | Baseline to Week 52
  BMD of the LS is measured using DEXA

SECONDARY OUTCOMES:
All Participants: Change From Baseline to Weeks 24, 52, and 104 in LS BMD Z-score Measured by DEXA | Baseline to Week 24, Week 52 and Week 104
Group 2: Change From Baseline to Weeks 24 and 104 in LS BMD Z-score Measured by DEXA | Baseline to Week 24 and Week 104
Group 2: Change From Baseline to Weeks 24, 52 and 104 in Total Body Less Head Bone Mineral Density (TBLH BMD) Z-score Measured by DEXA | Baseline to Week 24, Week 52 and Week 104
Group 2: Change From Baseline to Weeks 24, 52 and 104 in Total Hip BMD Z-score Measured by DEXA | Baseline to Week 24, Week 52 and Week 104
Group 2: Change From Baseline to Weeks 12, 24 and 52 in Circulating Bone Metabolism Biomarkers | Baseline to Week 12, Week 24 and Week 52
  Bone biomarkers are produced from the bone remodeling process and include bone formation biomarkers, bone resorption biomarkers and regulators of bone turnover.
All Participants: Change From Baseline to Weeks 12, 24 and 52 in Circulating Bone Metabolism Biomarkers | Baseline to Week 12, Week 24, and Week 52
  Bone biomarkers are produced from the bone remodeling process and include bone formation biomarkers, bone resorption biomarkers and regulators of bone turnover.
All Participants: Mean Number Per Participants of New Low-trauma Long-bone or Vertebral Fractures (VF) | Baseline to Week 52 and Week 104
  "A low-trauma fracture is defined as one occurring spontaneously or resulting from a fall from a standing height or less, without major trauma or the influence of an external force (e.g. motor vehicle accident)".
All Participants: Percentage of Participants With New Low-trauma Long-bone or VF | Baseline to Week 52 and Week 104
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to approximately 30 Months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant temporally associated with the use of a study treatment, whether or not considered related to the study treatment
Percentage of Participants With Serious Adverse Events (SAEs) | Up to approximately 30 Months
  A SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability or incapacity; is a congenital anomaly or birth defect; medically significant.
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Up to approximately 30 Months
Observed Serum Concentration of Satralizumab at Specified Trough Timepoints up to Week 104 | Up to Week 104
Apparent Clearance of Satralizumab | Up to Week 104
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution of Satralizumab | Up to Week 104
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Area Under the Concentration-time Curve of Satralizumab | Up to Week 104
  Area under the concentration-time curve from time zero to the last quantifiable concentration of Satralizumab in plasma.
Percentage of Participants With Anti-drug Antibodies (ADAs) at Baseline and During the Study | Up to approximately 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (9):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California Davis Medical Center, Sacramento, California
  - Children's Healthcare of Atlanta Center for Advanced Pediatrics, Atlanta, Georgia
  - University of Massachusetts Memorial Childrens Medical Center, Worcester, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Billings Clinic Research Center, Billings, Montana
  - Columbia University Medical Center, New York, New York
  - Neurology Rare Disease Center, Flower Mound, Texas
  - Child's Hosp King's Daughters, Norfolk, Virginia
- Rigshospitalet;Klinik for Børn og Unge med Hjerne- og Nervesygdomme, København Ø, Denmark
- Italy (3):
  - Policlinico Agostino Gemelli, Rome, Lazio
  - IRCCS Istituto G. Gaslini, Genoa, Liguria
  - Fondazione IRCCS Istituto Neurologico ?Carlo Besta?, Milan, Lombardy
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
  - Uniwersyteckie Centrum Kliniczne WUM, Centralny Szpital Kliniczny, Warsaw
- Spain (4):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital U. Central de Asturias, Asturias, Principality of Asturias
  - Hospital Universitario Torrecardenas;Servicio de Neurologia, Almería
  - Hospital Universitario la Fe, Valencia
- Ukraine (4):
  - Ivano-Frankivsk Regional Children Clinical Hospital, Ivano-Frankivsk, Kharkiv Governorate
  - Ukrainian medical rehabilitation center for children with organic lesions of the nervous system, Kyiv, KIEV Governorate
  - Ohmatdyt - National Specialized children's hospital of MoH of Ukraine, Kyiv
  - Lvivska oblasna tsentralna likarnia, Lviv

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing